CLINICAL TRIAL: NCT00247260
Title: A Study of the Safety Profile of Three Escalating Radioactivity Levels of 32P BioSilicon Delivered With the SIMPL Needle as Intratumoural Implantations in Patients With Unresectable Hepatocellular Carcinoma
Brief Title: Safety of 32P BioSilicon in Patients With Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: pSiVida Limited (Industry)
Collaborators: pSiOncology Private Limited (Unknown)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIOSP 202; NCT00252265 (obsolete NCT alias)
Record Dates: First submitted 2005-10-31; First posted 2005-11-01 (Estimated); Last update posted 2007-03-15 (Estimated); Status verified 2005-10

CONDITIONS: Liver Cancer
Keywords: HCC; Primary Liver Cancer
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular

INTERVENTIONS:
Device: 32P BioSilicon

SUMMARY:
Brachytherapy is a recent technique used in the treatment of tumours and involves the use of radioactive sources brought into close contact with the target tissues. One of the principal benefits of brachytherapy is that high radiation doses can be localised within the tumour with the consequence of minimal side effects. 32P is a radionuclide ideal for brachytherapy as it has high energy beta emitting properties, typically a maximum tissue range of about 8 mm and a half life of 14.3 days. 32P BioSiliconTM is an active implantable medical device encapsulating 32P within the internal microcrystalline structure of highly pure inert silicon and acts as a sealed source for the provision of 32 phosphorous.

Tumours targeted with 32P BioSiliconTM are hypothesized to show a reduction in volume with a low incidence of side effects associated with the treatment. Prolongation of survival and improved quality of life would be favourable outcomes of the investigational product.

DETAILED DESCRIPTION:
The study will enroll between 48 to 50 patients from all sites. Patients will be enrolled sequentially into the three groups, starting wth Group 1 which will investigate the lower radioactivity level and then progress to a higher radioactivity level in Group 2 and then Group 3. The approval to enrol patients into the next group will be assessed and determined by a Data Monitoring Board. All patients will be followed up to 52 weeks from the start date of primary implantations.

Patients will receive intratumoural implantations of 32P BioSiliconTM under imaging guidance and local anaesthesia by designated interventional radiologists, using the SIMPL needle or conventional needles depending on the size and location of the tumour as assessed by the designated interventional radiologists. There are only a designated number of sites that will perform the implantation procedure although there are multiple sites recruiting and following up with patients.

* Tumour assessment, tumour calculation and measurement will be performed by an independent radiologist. CT scans from all participating sites will be sent in DICOM format to the designated radiologist for assessment.
* Safety assessment and grading of CTCAE will be performed by the same investigator for that same patient throughout the entire study period. There will be an interim analysis when all patients complete 24 weeks evaluating the safety profile and target tumour response of the patients.
* 32P BioSiliconTM will be prepared by designated personnel licensed to handle radioactive products and all radioactive waste will be handed and managed as per the institution's guidelines and in compliance with local regulatory requirements.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent.
2. Male or female patients equal to or greater than 18 years old.
3. Patients with diagnosis of hepatocellular carcinoma (HCC) meeting one of the criteria below:

   1. Histology OR
   2. Radiological evidence'*' of HCC demonstrated by dynamic contrast enhanced computed tomography (CT) or dynamic contrast enhanced magnetic resonance imaging (MRI) >/ 1cm AND serum AFP of at least 400 mcg/L OR
   3. Radiological evidence'*' of HCC demonstrated by dynamic contrast CT or dynamic contrast enhanced MRI >/ 1cm AND serology positive for hepatitis B or C infection.

   '*' Criteria for radiological evidence of HCC are: central enhancement on hepatic arterial phase AND wash out on portal venous or delayed phase.
4. Hepatic tumour mass not amenable to surgical resection or patient refuses surgery.
5. ECOG performance status 0 - 2.
6. Okuda stage I - II
7. Total volume of any single treatable tumour not more than 65 cc (not more than approximately 5 cm in longest dimension).
8. Total treatable volume of not more than 125 cc (Group 1), 111 cc (Group 2), 139 cc (Group 3) - as defined by maximum radioactivity level (MBq) for the respective groups.
9. Adequate haematological, renal and hepatic functions as defined by the following laboratory values obtained within 14 days prior to Visit 2

   * Absolute granulocyte count (AGC) >/1500 cells/mm3
   * Serum creatinine < 2 times upper limit of normal (ULN)
   * Serum bilirubin < 3 times ULN
   * ALT (SGPT) < 5 times ULN and/or AST (SGOT) < 5 times ULN within 24 hours prior to implantation (Supportive care and correction permitted) Platelet count >/ 60,000/mm3 (60 x 10^9/L)
   * Prothrombin time < 3 seconds prolonged
10. Women of childbearing potential must have a negative urine pregnancy test within three days of Visit 2.
11. Contraception must be used (both male and female) for six months after implantation and during the duration of the whole study.
12. Patients must be accessible for treatment and follow up.

Exclusion Criteria:

1. Clinical encephalopathy
2. Patients younger than 18 years old.
3. No life threatening tumours in other sites (e.g. brain)
4. Less than four weeks after local therapy with radiofrequency ablation (RFA), or ethanol, and less than six weeks after local therapy with transarterial chemoembolization therapy (TACE), or since prior chemotherapy or biologic therapy (e.g. immunotherapy, systemic vaccine therapy).
5. Prior radiotherapy to liver, pancreas or gastrointestinal tract.
6. Total volume for each tumour is greater than 65 cc (greater than approximately 5 cm in longest dimension).
7. Amenable to surgery.
8. Pregnant or lactating females.
9. Other diagnosed malignancy within the last five years, which may impact on study outcome.
10. Life expectancy of less than 12 weeks.
11. Patients with a significant history of cardiac disease, that is, uncontrolled high blood pressure, unstable angina, congestive heart failure, myocardial infarction within the past three months and cardiac ventricular arrhythmias requiring medication.
12. Patients with serious active infection or other serious underlying medical conditions that would impair the ability of the patient to receive protocol treatment at implantation visits.
13. Patients with any condition (e.g. psychological) that does not permit compliance with the protocol.
14. Patients who are known to be HIV positive. Testing is not required in the absence of clinical signs and symptoms suggestive of HIV infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2005-10; Study Completion 2007-02

PRIMARY OUTCOMES:
This is a multicentre, open label study to evaluate the safety and efficacy of three escalating radioactivity levels (MBq) of 32P BioSiliconTM in patients with unresectable hepatocellular carcinoma

SECONDARY OUTCOMES:
To evaluate the safety profile of three escalating radioactivity levels (MBq) of 32P BioSiliconTM given as intratumoural implantations in patients with unresectable hepatocellular carcinoma
To evaluate the systemic distribution of 32P BioSiliconTM and soluble P32, following the intratumoural implantations
To evaluate the safety and performance of the SIMPLTM needle
To evaluate the target tumour response of three escalating radioactivity levels (MBq) of 32P BioSiliconTM
To evaluate the duration of target tumour response and overall survival rates
To evaluate the association between tumour marker serum alpha-fetoprotein (AFP) and target tumour response with the three radioactivity levels (MBq)

CONTACTS AND LOCATIONS:
Overall Officials: Pierce Chow, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Outram Road, Singapore

REFERENCES:
- See also: BrachySil A Novel Targeted Cancer Therapy — http://www.psivida.com